CLINICAL TRIAL: NCT02269319
Title: A Phase 2, Multicenter, Randomized, Double-blind Study to Evaluate the Safety and Efficacy of MRX-I Versus Linezolid in Adult Subjects With Acute Bacterial Skin and Skin Structure Infection
Brief Title: MRX-I Versus Linezolid for the Treatment of Acute Bacterial Skin and Skin Structure Infection
Acronym: ABSSSI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MicuRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRX-I-03
Record Dates: First submitted 2014-10-11; First posted 2014-10-21 (Estimated); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2017-01

CONDITIONS: Bacterial Infections
Keywords: ABSSSI; MRX-I; Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRX-I (Experimental): MRX-I tablets 800 mg given twice a day for 10 days
  Interventions: Drug: MRX-I
- Linezolid (Active Comparator): Linezolid 600 mg given twice a day for 10 days
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: MRX-I — Oral MRX-I 800mg given twice a day for 10 days
  Arms: MRX-I
Drug: Linezolid — Oral linezolid 600mg given twice a day for 10 days
  Other Names: Zyvox
  Arms: Linezolid

SUMMARY:
The purpose of this study is to determine whether MRX-I is as safe and effective as Linezolid in the treatment of adult patients with acute bacterial skin and skin structure infections

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic signs of infection diagnosed with acute bacterial skin and skin structure infection (ABSSSI)
* Diagnosed with Cellulitis/ erysipelas, major cutaneous abscess, or wound infections

Exclusion Criteria:

* Uncomplicated skin infections
* Severe sepsis or septic shock
* ABSSSI solely due to gram-negative pathogens
* Prior systemic antibiotics within 96 hours of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRX-I | Linezolid
Started | 80 | 40
Completed | 75 | 36
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 4 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Instructions not followed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRX-I | Linezolid | Total
Number analyzed (Participants) | 80 | 40 | 120
Age, Continuous [Mean (Full Range); unit: years] | 37.9 [20 to 62] | 38.8 [22 to 61] | 38.2 [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 13 | 40
  Male | 53 | 27 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients at the Early Assessment Visit With a 20% Reduction in ABSSSI Lesion Size Compared to Baseline
Description: * Did not receive a systemic antibacterial agent with activity against gram-positive organisms
  * Did not die of any cause up to EA
Time Frame: 48-72 hours
Population: Intent-to-Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | MRX-I | Linezolid
Number analyzed (Participants) | 80 | 40
Participants | 72 | 35

2. Secondary Outcome: Number of Patients at EOT With a 80% Reduction in ABSSSI Lesion Size Compared to Baseline
Time Frame: Day 10
Population: Intent-to-Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | MRX-I | Linezolid
Number analyzed (Participants) | 80 | 40
Participants | 70 | 32

ADVERSE EVENTS:
Time Frame: 39 days
Arm/Group | MRX-I | Linezolid
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/80 | 0/40
Other Adverse Events (participants affected / at risk) | 47/80 | 12/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRX-I (N=80) | Linezolid (N=40)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) — Moderate SAE unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MRX-I (N=80) | Linezolid (N=40)
Nausea (Gastrointestinal disorders) | 12 | 4
Abscess (Infections and infestations) | 9 | 3
Vomiting (Gastrointestinal disorders) | 7 | 3
Cellulitis (Skin and subcutaneous tissue disorders) | 5 | 1
Urinary Tract Infection (Infections and infestations) | 5 | 0
Hypertension (Vascular disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 0
Upper Respiratory Tract Infections (Infections and infestations) | 3 | 0

LIMITATIONS AND CAVEATS:
Proof of concept study was limited in size and scope. Given the number of male to female subjects, the interpretation of the results were limited. Since the duration of therapy was up to 10 days, assessment of long-term safety risks was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes